CLINICAL TRIAL: NCT02544321
Title: Bromocriptine Quick Release (QR) as Adjunct Therapy in Type 1 Diabetes
Brief Title: Bromocriptine Quick Release (BCQR) as Adjunct Therapy in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-1309; UL1TR001082 (NIH)
Record Dates: First submitted 2015-08-26; First posted 2015-09-09 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Bromocriptine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromocriptine QR (Active Comparator): 4 weeks of investigational drug Bromocriptine QR
  Interventions: Drug: Bromocriptine
- Placebo (Placebo Comparator): 4 weeks of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bromocriptine
  Other Names: Bromocriptine Quick Release (BCQR)
  Arms: Bromocriptine QR
Other: Placebo
  Arms: Placebo

SUMMARY:
Type 1 diabetes (T1D) continues to be a disease plagued by hyperglycemia, insulin resistance (IR), and increased cardiovascular disease (CVD) despite advances in insulin delivery and glucose monitoring. Therefore new approaches are needed. Bromocriptine (BC), a dopamine (DA) agonist, has long been widely used for treating Parkinson's disease and prolactinoma. Its recent approval in a quick release formulation, BCQR, for type 2 diabetes (T2D) is an exciting development, representing a novel mechanism for improving IR. BCQR has not been studied in T1D, but it's mechanism of action, mechanistic studies, and preliminary data support the proposed study of possible benefits of BCQR on insulin action, glycemic control, and the vasculature in T1D. This study has received an exemption from the FDA to study BCQR in adults with T1D and an IND approval (131360) to study BCQR in adolescents with T1D. This is a random-order, double-blind, placebo-controlled study of a 4 week intervention. Outcomes will include fasting and postprandial glucose, glycemic variability, insulin dosing, hypoglycemia frequency and awareness, sleep quality, and metabolic hormone levels.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes (T1D) of >1 year duration based on a clinical course consistent with T1D and rapid conversion to insulin requirement after diagnosis.
2. HbA1c 6.5-10% (adults) or any HbA1c up to 12% (pediatrics)
3. age 12-60 years of age

Exclusion Criteria:

1. Any comorbid condition associated with inflammation, insulin resistance, or dyslipidemia including cancer, heart failure, active or end stage liver disease, kidney disease (except microalbuminuria), inadequately treated thyroid disease, or rheumatologic disease;
2. Tobacco or marijuana use;
3. Pregnancy;
4. Regular or frequent oral steroid use;
5. Current use of insulin sensitizing medications, neuroleptics, ergot-related medications, or triptan medications for migraine,
6. Diagnosis or history of psychosis,
7. Diabetes of other cause such as Maturity Onset Diabetes of the Young or cystic fibrosis-related diabetes.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2015-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Schauer, MD, PhD, Principal Investigator — University of Colorado, Denver; Kristen Nadeau, MD, MS, Principal Investigator — Children's Hospital Colorado/University of Colorado
Locations (1):
- University of Colorado-Denver, Anshutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Tell SS, Schafer M, Vigers T, Baumgartner AD, Lyon E, Gross S, Polsky S, Snell-Bergeon JK, Schauer IE, Nadeau KJ. Bromocriptine quick-release as adjunct therapy in youth and adults with type 1 diabetes: A randomized, placebo-controlled crossover study. Diabetes Obes Metab. 2022 Nov;24(11):2148-2158. doi: 10.1111/dom.14800. Epub 2022 Jul 25. PMID 35712800

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants screen failed or withdrew from the study after enrollment, but prior to starting the study.
Groups:
- Bromocriptine QR, Then Placebo: 4 weeks of investigational drug Bromocriptine QR, then 4 weeks of placebo.
- Placebo, Then Bromocriptine QR: 4 weeks of placebo, then 4 weeks of investigational drug Bromocriptine QR
Period: Overall Study
Arm/Group | Bromocriptine QR, Then Placebo | Placebo, Then Bromocriptine QR
Started | 43 | 43
Completed First Treatment | 43 | 41
Completed Washout | 43 | 41
Started Second Treatment | 42 | 40
Completed | 41 | 39
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes all subjects who completed at least one phase of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromocriptine QR, Then Placebo | Placebo, Then Bromocriptine QR | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Adults and adolescents are divided by rows
  years
    Adults: number analyzed (Participants) | 21 | 21 | 42
    Adults | 44.1 (9.0) | 38 (10.0) | 41.1 (9.9)
    Adolescents: number analyzed (Participants) | 22 | 20 | 42
    Adolescents | 16.5 (2.8) | 15.6 (2.7) | 16.1 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Adults and adolescents are divided by rows
  Participants
    Adults: number analyzed (Participants) | 21 | 21 | 42
    Adults: Female | 12 | 11 | 23
    Adults: Male | 9 | 10 | 19
    Adolescents: number analyzed (Participants) | 22 | 20 | 42
    Adolescents: Female | 15 | 9 | 24
    Adolescents: Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adults and adolescents are divided by rows
  Participants
    Adults: number analyzed (Participants) | 21 | 21 | 42
    Adults: Hispanic or Latino | 0 | 1 | 1
    Adults: Not Hispanic or Latino | 21 | 20 | 41
    Adults: Unknown or Not Reported | 0 | 0 | 0
    Adolescents: number analyzed (Participants) | 22 | 20 | 42
    Adolescents: Hispanic or Latino | 1 | 2 | 3
    Adolescents: Not Hispanic or Latino | 21 | 18 | 39
    Adolescents: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adults and adolescents are divided by rows
  Participants
    Adults: number analyzed (Participants) | 21 | 21 | 42
    Adults: American Indian or Alaska Native | 0 | 0 | 0
    Adults: Asian | 0 | 0 | 0
    Adults: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adults: Black or African American | 0 | 0 | 0
    Adults: White | 21 | 21 | 42
    Adults: More than one race | 0 | 0 | 0
    Adults: Unknown or Not Reported | 0 | 0 | 0
    Adolescents: number analyzed (Participants) | 22 | 20 | 42
    Adolescents: American Indian or Alaska Native | 0 | 0 | 0
    Adolescents: Asian | 0 | 0 | 0
    Adolescents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescents: Black or African American | 0 | 1 | 1
    Adolescents: White | 22 | 19 | 41
    Adolescents: More than one race | 0 | 0 | 0
    Adolescents: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 41 | 84

OUTCOME MEASURES:

1. Primary Outcome: Mean Glucose
Description: At the end of each 4 week intervention period, we will measure the effect of Bromocriptine Quick Release on average glucose levels (mg/dl) by continuous glucose monitoring
Time Frame: 4 weeks
Population: Data reflects average glucose levels.
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Groups:
- Bromocriptine QR (Adolescents); Bromocriptine QR (Adults): 4 weeks of investigational drug Bromocriptine QR
  Bromocriptine
- Placebo (Adolescents); Placebo (Adults): 4 weeks of placebo
  Placebo
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dl | 182 (5) | 165 (5) | 181 (5) | 165 (5)

2. Primary Outcome: Insulin Dosing
Description: At the end of each 4 week intervention period, we will measure the effect of BCQR on insulin dosing (units//kg/day)
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: units//kg/day
Groups:
- Bromocriptine QR (Adults): 4 weeks of investigational drug Bromocriptine QR
- Placebo (Adults): 4 weeks of placebo
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40 | 40 | 40
units//kg/day | 0.9 (.03) | 0.54 (.02) | 0.88 (.03) | 0.56 (0.02)

3. Primary Outcome: Brachial Artery Distensibility
Description: At the end of each 4 week intervention period, we will measure the brachial artery distensibility as a measure of vascular stiffness by Dynapulse (%/mmHg). A larger number indicates less stiffness (ie greater compliance).
Time Frame: 4 weeks
Population: Compared for placebo versus BCQR after 4 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: %/mmHg
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40 | 40 | 40
%/mmHg | 6.35 (0.19) | 6.2 (0.2) | 6.14 (0.19) | 6.4 (0.2)

4. Primary Outcome: Hyperemia Peripheral Arterial Tonometry (RH-PAT): Reactive Hyperemia Index (RHI)
Description: At the end of each 4 week intervention period, we will measure the reactive hyperemia Index (RHI). The Reactive Hyperemia Index (RHI) measures increased bloodflow after vascular occlusion. Higher scores indicate lower CVD risk and a better outcome, Scores of less than 1.67 may be considered abnormal. Scores of 1.67 1.67-2.09 may be considered borderline, and scores of 2.10 or higher my be considered normal.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40 | 40 | 40
score on a scale | 1.95 (0.09) | 2.1 (0.1) | 2.24 (0.09) | 2.2 (0.1)

5. Secondary Outcome: Mean Glycemic Variability
Description: At the end of each 4 week intervention period, we will measure the effect of Bromocriptine Quick Release on glycemic variability throughout the day (mg/dl), measured as SD of all glucose values throughout the last 7 days of intervention. Incorrectly initially entered as primary outcome. per protocol this has always been a secondary outcome.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dl | 71 (2.1) | 61 (2.5) | 73 (2.1) | 63 (2.5)

6. Secondary Outcome: Hypoglycemia Awareness
Description: At the end of each 4 week intervention period, we will measure Hypoglycemia Awareness using the Gold method (7 point Likert scale: Possible scores range from 1 to 7. higher scores indicate more impaired awareness of hypoglycemia, and a worse outcome), Clarke method (8 question questionnaire characterizing hypoglycemia awareness. Possible scores range from 0-7, with higher scores indicating less awareness and a worse outcome), and the McAuley score (list of symptoms with a 7 point Likert scale for each. Possible scores range from 1-7 for each item, and are averaged across all symptoms, for a total possible score range of 1-7, with higher scores indicating more symptom awareness, and a better outcome).
  Incorrectly initially entered as primary outcome. per protocol this has always been a secondary outcome.
Time Frame: 4 weeks
Population: Unadjusted least square means by mixed procedure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 41 | 41 | 41
score on a scale
  Gold method scores | 2.15 (1.31) | 3.02 (1.67) | 2.00 (1.18) | 3.15 (1.59)
  Clarke method scores | 1.36 (1.23) | 2.33 (1.90) | 1.33 (1.20) | 2.67 (1.84)
  McAuley score | 3.25 (0.22) | 3.40 (0.31) | 3.21 (0.22) | 2.90 (0.29)

7. Secondary Outcome: Augmentation Index
Description: At the end of each 4 week intervention period, the % will be measured by SyphgmoCor. The Augmentation Index measures vascular stiffness by comparing pulse pressure of the reflected wave to the primary wave. HIGHER scores indicate greater vascular stiffness and higher cardiovascular risk, but a normal range has not been clearly defined. Presented as AI normalized to a heart rate of 75 (AI75).
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of pressure wave
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40 | 40 | 40
Percentage of pressure wave | 10.42 (1.71) | -2.0 (1.8) | 12.52 (1.72) | -2.5 (1.8)

8. Secondary Outcome: Heart Rate Variability (Adults)
Description: At the end of each 4 week intervention period we will measure the autonomic function by ECG. Ratio of maximum heart rate/minimum heartrate during a valsalva maneuver.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Bromocriptine QR (Adults) | Placebo (Adults)
Number analyzed (Participants) | 40 | 40
ratio | 1.09 (0.05) | 1.14 (0.05)

9. Secondary Outcome: Heart Rate Variability (Adolescents)
Description: At the end of each 4 week intervention period we will measure the autonomic function by HRV measured by endopat and reported using the single gold standard measure of SDNN (standard deviation of beat to beat time interval). Normal is >100, 50-100 indicates compromised autonomic function.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Bromocriptine QR (Adolescents) | Placebo (Adolescents)
Number analyzed (Participants) | 40 | 40
milliseconds | 73 (5) | 76.4 (4.9)

10. Secondary Outcome: Sleep Duration
Description: At the end of each 4 week intervention period, measurements of sleep duration on weekdays and weekends (minutes) by a Philips Spectrum Plus sleep monitor will be obtained.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
minutes
  weekdays | 433 (69) | 394 (59) | 414 (47) | 402 (62)
  weekends | 486 (81) | 458 (95) | 464 (85) | 453 (98)

11. Secondary Outcome: Sleep Quality
Description: At the end of each 4 week intervention period, measurements of sleep efficiency (percent of time in bed spent asleep) during the week and on weekends by a Philips Spectrum Plus sleep monitor will be obtained.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
percent
  efficiency during the week | 87.9 (5.3) | 90.4 (4.2) | 89.0 (4.1) | 90.4 (4.4)
  efficiency weekends | 88.3 (4.8) | 89.7 (5.0) | 89.0 (5.4) | 90.9 (3.6)

12. Secondary Outcome: Metabolic Markers-glucose and Triglycerides
Description: At the end of each 4 week intervention period, glucose, insulin, triglycerides, NEFA, GLP-1, and glucagon area under the curve will be measured during Mixed Meal Tolerance Test.
Time Frame: 4 weeks
Population: glucose and triglyceride total AUC least square means +/- SD
Measure: Least Squares Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
mg*hr/dL
  Glucose | 11735 (7180) | 9228 (5530) | 11356 (5990) | 12357 (6962)
  Triglycerides | 3452 (2878) | 3445 (4582) | 3066 (2040) | 3460 (4634)

13. Secondary Outcome: Metabolic Markers-fatty Acids
Description: as for outcome 12
Time Frame: 4 weeks
Population: Non-esterified fatty acids total AUC least square means +/- SD
Measure: Least Squares Mean (Standard Deviation); unit: microEq*hr/L
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
microEq*hr/L | 123334 (115005) | 75561 (52616) | 93661 (58385) | 67497 (46017)

14. Secondary Outcome: Metabolic Markers-glucagon
Description: as for outcome 12
Time Frame: 4 weeks
Population: glucagon total AUC least square means +/- SE
Measure: Least Squares Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
pg*hr/mL | 2398 (1959) | 2160 (1361) | 2011 (1252) | 2350 (1491)

15. Secondary Outcome: Metabolic Markers - GLP1
Description: as for outcome 12
Time Frame: 4 weeks
Population: GLP-1 total AUC least square means +/- SD
Measure: Least Squares Mean (Standard Deviation); unit: pmol*hr/L
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
pmol*hr/L | 661 (435) | 872 (563) | 766 (392) | 1196 (728)

16. Secondary Outcome: Metabolic Markers - Insulin
Description: as for outcome 12
Time Frame: 4 weeks
Population: insulin total AUC least square means +/- SD
Measure: Least Squares Mean (Standard Deviation); unit: microIU*hr/mL
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
Number analyzed (Participants) | 42 | 42 | 42 | 42
microIU*hr/mL | 4162 (2496) | 2386 (1087) | 4001 (3209) | 2379 (1160)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Bromocriptine QR (Adolescents) | Bromocriptine QR (Adults) | Placebo (Adolescents) | Placebo (Adults)
All-Cause Mortality (participants affected / at risk) | 1/42 | 1/42 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 13/42 | 17/42 | 1/42 | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromocriptine QR (Adolescents) (N=42) | Bromocriptine QR (Adults) (N=42) | Placebo (Adolescents) (N=42) | Placebo (Adults) (N=42)
severe hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — participant had episode of severe hypoglycemia working at high altitude as a diabetes camp counselor without adjusting insulin dosing as instructed for the change in altitude/activity Event resolved without sequelae.
diagnosed with RA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bromocriptine QR (Adolescents) (N=42) | Bromocriptine QR (Adults) (N=42) | Placebo (Adolescents) (N=42) | Placebo (Adults) (N=42)
nausea (Gastrointestinal disorders) | 13 | 17 | 1 | 3 — shortly after dose. only caused one w/d.
orthostasis (Vascular disorders) | 4 | 6 | 0 | 2 — occurred shortly after dosing. not sever enough to cause d/c.
fatigue (General disorders) | 1 | 5 | 0 | 3
headache (General disorders) | 2 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT02544321/Prot_SAP_000.pdf